CLINICAL TRIAL: NCT02711787
Title: Efficacy of Short-Term Robot-Assisted Rehabilitation in Patients With Hand Paralysis After Stroke: a Randomized Clinical Trial
Brief Title: Efficacy of Robot-Assisted Rehabilitation of Hand Paralysis After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Project Code:RC-2015-Gloreha
Record Dates: First submitted 2016-03-05; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Stroke
Keywords: Hand; Paralysis; Stroke
MeSH Terms: conditions — Stroke; Paralysis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Robotic device Gloreha (Gloreha, Idrogenet, Italy) and traditional rehabilitation, 60-minute session for 3 consecutive weeks (3 days/week).
  Interventions: Device: Experimental group; Device: traditional rehabilitation
- Control group (Active Comparator): Physiotherapy, occupational therapy and traditional rehabilitation, 60-minute session for 3 consecutive weeks (3 days/week).
  Interventions: Device: Control group; Device: traditional rehabilitation

INTERVENTIONS:
Device: Experimental group — Robotic assisted passive mobilization (Gloreha, Idrogenet, Italy) and traditional rehabilitation.
  Arms: Experimental group
Device: Control group — Physiotherapy and occupational therapy.
  Arms: Control group
Device: traditional rehabilitation — Assisted stretching, shoulder and arm exercises, and functional reaching tasks

SUMMARY:
Among robotic devices, Gloreha, with its compliant mechanical transmission, may represent an easily applied innovative solution to rehabilitation, because the hand can perform grasp and release activities wearing the device by mean of a flexible and light orthosis. Our objective on this research was to the robotic assisted motion and activity in additional to physiotherapy (PT) and occupational therapy (OT), on stroke patients with hand paralysis.

DETAILED DESCRIPTION:
The investigators evaluated the effectiveness of a robotic-assisted motion and activity in additional to physiotherapy (PT) and occupational therapy (OT), on stroke patients with hand paralysis. A randomized controlled trial. The experimental group received a passive mobilization of the hand through the robotic device Gloreha and control group received a PT and OT for 3 consecutive weeks (3 days/week) in addition to traditional rehabilitation. Outcomes included the National Institutes of Health Stroke Scale (NIHSS), Modified Ashworth Scale (MAS), Barthel index (BI), Motricity index (MI), short version of the Disabilities of the Arm, Shoulder and Hand (quickDASH), and the Visual Analogue Scale (VAS) measurements. All measures were collected at baseline and end of the intervention (3 weeks).

ELIGIBILITY:
Inclusion Criteria:

* acute phase of stroke
* first stroke episode.
* no history of peripheral nerve injury or musculoskeletal disease
* no contracture of the affected wrist or fingers (Modified Ashworth<3)
* no history of any invasive procedure (Botulinum toxin type A) for the treatment of spasticity for at least 6 months prior to the start of this study.
* paralysis of the wrist and fingers

Exclusion Criteria:

* unstable medical disorders, active Complex Regional Pain Syndrome (CRPS) severe spatial neglect, aphasia, or cognitive problems.
* scored greater than 4 points on the Beck Depression Inventory (BDI)
* more than 30 points in the State Trait Anxiety Inventory (STAI)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from National Institutes of Health Stroke Scale (NIHSS) | baseline, immediately post-intervention (3 weeks).

SECONDARY OUTCOMES:
Change from Visual analogue scale (VAS) | baseline, immediately post-intervention (3 weeks).
Change from Barthel Index (BI) | baseline, immediately post-intervention (3 weeks).
Change from Modified Ashworth Scale (MAS) | baseline, immediately post-intervention
Change from Disabilities of the Arm, Shoulder and Hand (quickDASH) | baseline, immediately post-intervention (3 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: JORGE H VILLAFAÑE, PhD, Principal Investigator — IRCCS Don Gnocchi Foundation

IPD SHARING:
Plan to Share IPD: No